CLINICAL TRIAL: NCT05595200
Title: Prevalence, Phenotypes, Predictors and Prognostic Implication of Obstructive Sleep Apnea in Pulmonary Hypertension
Acronym: POSAPH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: SAPH
Record Dates: First submitted 2022-10-22; First posted 2022-10-26 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Sleep Apnea; Obstructive Sleep Apnea; Pulmonary Hypertension; Epidemiology; Predictor; Prognosis; Outcomes; Mortality
Keywords: Sleep Apnea; Pulmonary Hypertension; Obstructive Sleep Apnea; Hypoxemia; Prognosis; Prevalence; Predictor; Phenotype; Outcome
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Hypertension, Pulmonary; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: All subjects diagnosed with pulmonary hypertension by right heart catheterization agreeing to participate and meeting inclusion criteria but not meeting exclusion criteria
  Interventions: Diagnostic Test: Level III portable sleep study

INTERVENTIONS:
Diagnostic Test: Level III portable sleep study — Recruited patients will undergo an overnight cardiorespiratory study using a Level III portable device before hospital discharge

SUMMARY:
The investigators propose a prospective, observational study to determine the impact of OSA and associated physiological parameters on clinical outcomes in patients with pulmonary hypertension. The prevalence, phenotypes, and predictors of OSA in the setting of pulmonary hypertension will also be investigated. Adult patients diagnosed with pulmonary hypertension by right heart catheterization are eligible. Recruited patients will undergo an overnight cardiorespiratory study using a Level III portable device before hospital discharge. The cardiorespiratory tracings during sleep will be analyzed and audited by a certified sleep physician. The patients will be divided into two groups based on the apnea-hypopnea index (AHI): OSA (AHI ≥ 5) and non-OSA (AHI<5) groups. Hypoxemic parameters such as time percentage spent with oxygen saturation below 90% and nadir oxygen saturation were all collected. Baseline clinical characteristics, such as the Epworth sleepiness scales, were also obtained. The primary endpoint of this study was clinical worsening (CW), defined as the composite event of a reduction in exercise capacity, worsening in World Health Organization functional class, non-elective hospitalization for pulmonary hypertension, or all-cause mortality. Secondary endpoints include individual outcomes of clinical worsening and all-cause mortality.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a highly prevalent sleep-breathing disorder that affects over 1 billion adults worldwide, resulting in a substantial economic and medical burden. Multiple cardiovascular comorbidities and mortality are associated with OSA due to intermittent hypoxemia, intrathoracic pressure swings, sympathetic activation, endothelial dysfunction, and systemic inflammation. Large epidemiological studies have shown that OSA is more prevalent in patients with pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension than in the general population. Thus, elucidating the effects of OSA on adverse outcomes in patients with pulmonary hypertension is crucial in risk assessments and therapeutic recommendations for affected individuals. There is, however, insufficient evidence to determine whether OSA and associated physiological sequelae/phenotypes have a prognostic impact on these patients. The investigators propose a prospective, observational study to determine the impact of OSA and associated physiological parameters on clinical outcomes in patients with pulmonary hypertension. The prevalence, phenotypes, and predictors of OSA in the setting of pulmonary hypertension will also be investigated. Adult patients diagnosed with pulmonary hypertension by right heart catheterization are eligible. Recruited patients will undergo an overnight cardiorespiratory study using a Level III portable device before hospital discharge. The cardiorespiratory tracings during sleep will be analyzed and audited by a certified sleep physician. The patients will be divided into two groups based on the apnea-hypopnea index (AHI): OSA (AHI ≥ 5) and non-OSA (AHI<5) groups. Hypoxemic parameters such as time percentage spent with oxygen saturation below 90% and nadir oxygen saturation were all collected. Baseline clinical characteristics, such as the Epworth sleepiness scales, were also obtained. The primary endpoint of this study was clinical worsening (CW), defined as the composite event of a reduction in exercise capacity (15% compared with the previous six-minute walk distance), worsening in World Health Organization functional class, non-elective hospitalization for pulmonary hypertension (need for an intravenous diuretic or inotropic drugs, new targeted therapies, lung transplantation, or septostomy), or all-cause mortality. Secondary endpoints include individual outcomes of clinical worsening and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old
* Diagnosed with pulmonary hypertension by right heart catheterization

Exclusion Criteria:

* Pregnancy
* Central sleep apnea
* Previous treatment for sleep-disordered breathing
* Unavailable or incomplete sleep data
* Requiring nocturnal oxygen supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College diagnosed with pulmonary hypertension that meet inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical worsening | 1 year
  The composite event of a reduction in exercise capacity (15% compared with the previous six-minute walk distance), worsening in World Health Organization functional class, non-elective hospitalization for pulmonary hypertension (need for an intravenous diuretic or inotropic drugs, new targeted therapies, lung transplantation, or septostomy), or all-cause mortality.

SECONDARY OUTCOMES:
Individual clinical worsening outcomes | 1 year, 3 years and 5 years
  Number of patients with reduction in exercise capacity, reduction in WHO functional classes, non-elective hospitalization for pulmonary hypertension and all-cause mortality.
Clinical worsening | 3 year, 5 years
  The composite event of a reduction in exercise capacity (15% compared with the previous six-minute walk distance), worsening in World Health Organization functional class, non-elective hospitalization for pulmonary hypertension (need for an intravenous diuretic or inotropic drugs, new targeted therapies, lung transplantation, or septostomy), or all-cause mortality.
All-cause mortality | 1 year, 3 year, 5 years
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Center for Respiratory and Pulmonary Vascular Diseases, Fuwai hospital, CAMS & PUMC, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duan A, Huang Z, Hu M, Zhao Z, Zhao Q, Jin Q, Yan L, Zhang Y, Li X, An C, Luo Q, Liu Z. The comorbidity burden and disease phenotype in pre-capillary pulmonary hypertension: The contributing role of obstructive sleep apnea. Sleep Med. 2023 Jan;101:146-153. doi: 10.1016/j.sleep.2022.10.029. Epub 2022 Nov 2. PMID 36395719
- [Background] Huang Z, Duan A, Hu M, Zhao Z, Zhao Q, Yan L, Zhang Y, Li X, Jin Q, An C, Luo Q, Liu Z. Implication of prolonged nocturnal hypoxemia and obstructive sleep apnea for pulmonary hemodynamics in patients being evaluated for pulmonary hypertension: a retrospective study. J Clin Sleep Med. 2023 Feb 1;19(2):213-223. doi: 10.5664/jcsm.10286. PMID 36081323
- [Background] Hu M, Duan A, Huang Z, Zhao Z, Zhao Q, Yan L, Zhang Y, Li X, Jin Q, An C, Luo Q, Liu Z. Development and Validation of a Nomogram for Predicting Obstructive Sleep Apnea in Patients with Pulmonary Arterial Hypertension. Nat Sci Sleep. 2022 Aug 9;14:1375-1386. doi: 10.2147/NSS.S372447. eCollection 2022. PMID 35971464
- [Background] Huang Z, Duan A, Zhao Z, Zhao Q, Zhang Y, Li X, Zhang S, Gao L, An C, Luo Q, Liu Z. Sleep-disordered breathing patterns and prognosis in pulmonary arterial hypertension: A cluster analysis of nocturnal cardiorespiratory signals. Sleep Med. 2024 Jan;113:61-69. doi: 10.1016/j.sleep.2023.11.016. Epub 2023 Nov 13. PMID 37984019